CLINICAL TRIAL: NCT06111482
Title: Clinical Study to Evaluate Different Energy-based Devices for Aesthetic Treatments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EUN-PL01-2023
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Dermatologic Conditions
MeSH Terms: interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Intervention Model Description: Subjects will be treated with an intended pulsed light device. Subjects may also receive split treatments where one side of the face and/or body will be treated with the study device, and the contralateral side will be treated with a similar IPL device or a similar microneedling device. Randomization will not be used as the group the subject will be assigned to will be determined based on dermatologic condition the subject presents with and this will be determined by the Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- IPL only (Experimental): Group A will be treated with an intense pulsed light (IPL) device only. They may also receive split treatments where one side of the face and/or body will be treated with the study device and the contralateral side will be treated with a similar IPL device that is cleared for use by the FDA.
  Interventions: Device: Intense pulsed light.
- RF Microneedling Only (Experimental): Group B will be treated with a radiofrequency (RF) microneedling device only. They may also receive split treatments where one side of the face and/or body will be treated with the study device and the contralateral side will be treated with a similar RF microneedling device that is cleared for use by the FDA.
  Interventions: Device: Radiofrequency microneedling device
- RF Only (Experimental): Group C will be treated with an RF device only. They may also receive split treatments where one side of the face and/or body will be treated with the study device and the contralateral side will be treated with a similar RF device that is cleared for use by the FDA.
  Interventions: Device: Radiofrequency device
- Combination (Experimental): Group D will receive combination treatments and will be treated with 2 or more of the study devices.
  Interventions: Device: Intense pulsed light.; Device: Radiofrequency microneedling device; Device: Radiofrequency device; Device: Combined energy devices

INTERVENTIONS:
Device: Intense pulsed light. — The intense pulsed light (IPL) will be used for treating unwanted dermatologic conditions which may be on multiple areas of the body such as, but not limited to, the face, décolletage, back, legs, arms, and hands.
  Arms: Combination; IPL only
Device: Radiofrequency microneedling device — The microneedling device will be used for treating unwanted dermatologic conditions which may be on multiple areas of the body such as, but not limited to, the face, décolletage, back, legs, arms, and hands.
  Arms: Combination; RF Microneedling Only
Device: Radiofrequency device — The radio frequency device will be used for treating unwanted dermatologic conditions which may be on multiple areas of the body such as, but not limited to, the face, décolletage, back, legs, arms, and hands.
  Arms: Combination; RF Only
Device: Combined energy devices — The combined energy devices will be used for treating unwanted dermatologic conditions which may be on multiple areas of the body such as, but not limited to, the face, décolletage, back, legs, arms, and hands.
  Arms: Combination

SUMMARY:
The goal of the energy-based devices used in this study is to evaluate their safety and performance to treat unwanted dermatologic conditions.

DETAILED DESCRIPTION:
Up to 50 subjects will be enrolled at 1 study center. Subjects will be enrolled into 4 groups: Group A, Group B, Group C, or Group D. Subjects may enroll in more than one group, however the last treatment in the previous group would be at least 30 days before the subject is enroll in the next group if treatment area is the same.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 22 years of age or older.
* Willing to undergo at least 1 treatment with the study device(s).
* Understands and accepts obligation not to receive any other procedures in the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document

Exclusion Criteria:

* Is female and pregnant, has been pregnant within the last 3 months, is currently breast feeding or planning a pregnancy during the study period.
* Takes or has taken oral isotretinoin, such as Accutane®, within the last six months.
* Is using systemic steroids (e.g., prednisone, dexamethasone) prior to or during the course of treatment.
* Is receiving or has received gold therapy.
* Is taking medications that alter the wound-healing response or has a history of healing problems.
* Has an active localized or systemic infection, or an open wound in area being treated.
* Has a significant systemic illness, such as lupus, or an illness localized in area being treated.
* Has a seizure disorders triggered by light.
* Has a history of skin photosensitivity disorders.
* Has a history of hypertrophic scars or keloid formation.
* Has a history of radiation therapy in area to be treated.
* Received fillers or neurotoxin injections in the treatment area within the past 2 weeks.
* Has had a chemical or mechanical epilation within the last six weeks.
* Currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within the area to be treated 6 months to entering this study.
* Has any condition or is in a situation which in the investigator's opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.

Radiofrequency Device Only:

* Has a Pacemaker
* Has any embedded electronic devices that give or receive a signal.
* Has electronic implants, such as Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant.
* Is allergic to adhesives such as glues on medical tape: they should be alerted that a rash may occur on the neutral electronic monitoring pad (NEM or neutral pad) site, and an over-the-counter preparation may be used to treat the area.
* Has nerve insensitivity to heat in the treatment area or in the neutral pad placement area.
* Is allergic to topical anesthetic

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Maximum pain reported during treatment. | procedure (during device treatment)]
  The maximum pain during treatment per each device will be reported on a scale of 0(none) to 10 (maximum intolerable pain). This pain is recorded during when the patient is actively treated (when the patient comes in and receives a treatment from the device).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Doherty, Principal Investigator — Cynosure, LLC
Locations (1):
- Cynosure, Westford, Massachusetts, United States